CLINICAL TRIAL: NCT03586167
Title: Clinical Performance of a Monthly Replacement Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLY935-C004
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID014341 (Experimental): LID014341 contact lenses worn bilaterally (in both eyes) for 30 days on a daily wear basis
  Interventions: Device: LID014341 contact lenses
- Biofinity (Active Comparator): Comfilcon A contact lenses worn bilaterally for 30 days on a daily wear basis
  Interventions: Device: Comfilcon A contact lenses

INTERVENTIONS:
Device: LID014341 contact lenses — Investigational monthly replacement silicone hydrogel contact lenses with water gradient coating
  Arms: LID014341
Device: Comfilcon A contact lenses — Silicone hydrogel contact lenses
  Other Names: BIOFINITY©
  Arms: Biofinity

SUMMARY:
The purpose of this study is to assess the clinical performance of an investigational, coated silicone hydrogel contact lens over approximately 30 days of daily wear.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an informed consent form approved by an Institutional review board (IRB);
* Successful wear of spherical monthly replacement soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Best-corrected visual acuity (BCVA) 20/25 or better in each eye;
* Willing to stop wearing habitual contact lenses for the duration of study participation.

Exclusion Criteria:

* Any conditions or use of medications that could contraindicate contact lens wear;
* History of or plan to have refractive surgery in either eye;
* Irregular cornea in either eye;
* Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study;
* Current or history of intolerance, hypersensitivity or allergy to any component of the study products;
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Use of topical ocular medications and artificial tear or rewetting drops requiring instillation during contact lens wear;
* Habitual Biofinity contact lens wearers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (4):
- United States (4):
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Johns Creek, Georgia
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 study centers located in the US.
Pre-assignment Details: Of the 88 enrolled, 2 subjects exited as screen failures prior to randomization. This reporting group includes all randomized subjects (86).
Units Other Than Participants: eyes
Groups:
- LID014341: LID014341 contact lenses were worn bilaterally (in both eyes) for 30 days on a daily wear basis
- Biofinity: Comfilcon A contact lenses were worn bilaterally for 30 days on a daily wear basis
Period: Overall Study
Arm/Group | LID014341 | Biofinity
Started (Randomized and Treated) | 58; 116 eyes | 28; 56 eyes
Completed | 57; 114 eyes | 28; 56 eyes
Not Completed | 1; 2 eyes | 0; 0 eyes
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population included all subjects/eyes exposed to any study lens evaluated in this study (Safety Analysis Set).
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | LID014341 | Biofinity | Total
Number analyzed (Participants) | 58 | 28 | 86
Number analyzed (Eyes) | 116 | 56 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.6) | 40.7 (12.9) | 39.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 20 | 58
  Male | 20 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 56 | 26 | 82
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 52 | 25 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA)
Description: VA was tested monocularly (each eye individually) without visual correction under photopic (well-lit) conditions. VA was measured in logMAR (logarithm of the minimum angle of resolution), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. A lower numeric value represents better visual acuity. Both eyes contributed to the analysis. No formal statistical hypothesis testing was planned.
Time Frame: Day 30
Population: Safety Analysis Set. Overall number of units analyzed is the number of eyes with non-missing response.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | LID014341 | Biofinity
Number analyzed (Participants) | 57 | 28
Number analyzed (Eyes) | 114 | 56
logMAR | -0.09 (0.07) | -0.09 (0.07)

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 1 month (30 days)
Description: Adverse Event (AE) was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. This analysis population included all subjects/eyes exposed to any study lens evaluated in this study (Safety Analysis Set), based on treatment-specific exposure.
Arm/Group | LID014341 | Biofinity
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/28
Other Adverse Events (participants affected / at risk) | 0/58 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03586167/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03586167/SAP_001.pdf